CLINICAL TRIAL: NCT05256953
Title: Effect of Bilateral Erector Spinae Plan Block in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Yasemin Burcu Ustun, Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRCESP140619
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Pain, Postoperative
Keywords: Regional anesthesia; Erector spinae plane block; Post-operative analgesia; Laparoscopy; Open surgery; Colorectal surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Our study is a single center, prospective, randomized controlled, single-blinded, parallel group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients were randomly divided into two groups of 30 patients each. In the system where computer generated random numbers (SPSS v23.0, IBM, NewYork, USA) were used, ESP and GA groups were determined at a ratio of 1:1. Sealed and sequentially numbered envelopes were created. One hour before the operation, an experienced anesthesiologist, who was not involved in the intraoperative and postoperative follow-up of the patient and would only perform the block procedure, opened a sealed opaque sealed envelope to learn the group that the patient would be included in. There were two different physicians who performed intraoperative and postoperative follow-up. Both of the follow-up physicians were blind to the patient group. The care provider and investigator were also blinded to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP (Active Comparator): bilateral ESPB (total of 40 ml, %0.25 bupivacaine) + IV morphine PCA
  Interventions: Procedure: Erector spina plane block + general anesthesia
- Group GA (Active Comparator): only IV morphine PCA
  Interventions: Procedure: Only general anesthesia

INTERVENTIONS:
Procedure: Erector spina plane block + general anesthesia — Bilateral-injection ultrasound-guided bilateral erector spinae plane block
  Pre-operatively, with the patient in the sitting position, 20ml 0.25% bupivacaine will be administered between the T9 spinous process and the erector spinae muscles with the guidance of an ultrasound probe placed on a parasagittal plane. The same procedure was applied bilaterally.
  Intraoperative analgesia: After anesthesia induction tenoxicam 20 mg IV and 30 min. before the end of the surgery paracetamol (1gr) iv was applied.
  Postoperative analgesia: IV-PCA: The requested dose will be 20µg/kg morphine, the lock-in time will be 6-10 minutes, the 4-hour limit will be 80% of the total calculated dose.
  Rescue analgesia was provided with iv tramadol 30 mg boluses whenever the Visual analog scale pain score >3, (max doses 300 mg/day).
  Other Names: Group ESP
  Arms: Group ESP
Procedure: Only general anesthesia — Intraoperative analgesia: After anesthesia induction tenoxicam 20 mg IV and 30 min. before the end of the surgery paracetamol (1gr) iv was applied.
  Postoperative analgesia: IV-PCA: The requested dose will be 20µg/kg morphine, the lock-in time will be 6-10 minutes, the 4-hour limit will be 80% of the total calculated dose.
  Rescue analgesia was provided with iv tramadol 30 mg boluses whenever the Visual analog scale pain score >3, (max doses 300 mg/day).
  Other Names: Group GA
  Arms: Group GA

SUMMARY:
In this study, it was aimed to evaluate the effects erector spina plane block (ESPB) on postoperative opioid consumption in the first 24 hours and pain scores after colorectal surgery.

DETAILED DESCRIPTION:
Colorectal surgery can be applied for many reasons, among these reasons, colorectal cancer (CRC) takes the first place. With the understanding of the pathophysiological effects of analgesics better, the use of regional techniques in providing analgesia for patients undergoing colorectal cancer surgery has come to the fore. Depending on the surgical procedure, pain faced by patients is an important problem that must be deal with in the postoperative period.

In this study, the hypothesis was determined as "Pre-operatively, erector spina plane block (ESPB) performed as part of multimodal analgesia reduces postoperative morphine consumption and pain scores."

The patients were divided into two groups :

Group ESP (erector spinae plan):

In this group, patients will be administered bilateral ESPB (total of 40 ml, %0.25 bupivacaine) in addition to IV morphine patient-controlled analgesia (PCA) for the first 24 postoperative hours.

Group GA (general anesthesia):

In this group, patients will be administered only IV morphine patient-controlled analgesia (PCA) for the first 24 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years
* ASA I , II patients
* BMI<35 kg/m2 (body weight <100 kg , >45 kg)
* Patients who underwent colorectal surgery

Exclusion Criteria:

* Patients who underwent abdominoperineal resection
* Patients who were evaluated as unsuccessful block in the dermatomal examination performed after the block was applied.
* Patients diagnosed with OSAS
* Pregnancy and breastfeeding
* Contraindication of regional anesthesia (coagulopathy, abnormal INR, thrombocytopenia, infection at the injection site)
* Hypersensitivity to local anesthetics or a history of allergy
* Patients with a history of opioid use longer than four weeks
* Patients with severe psychiatric diseases such as psychosis or dementia that limit cooperation with the patient.
* Patients with anatomic deformity ( advanced scoliosis and kyphotic patients. Patients with pectus carinatum and pectus excavatum-like chest deformity )
* Patients who do not want to participate
* Patients who have had previous colorectal surgery, excluding diagnostic biopsies
* Patients who could not be reached by phone to inquire about their pain score at 3rd month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption in the first 24 hours | Postoperative day 1
  Morphine consumption in the first 24 hours were measured. Patients will be able to request opioids via a PCA device when their VAS score is above 3 at rest and during activity (coughing and deep breathing).

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative month 3
  Pain status at rest and while activity (coughing and deep breathing) were assessed by VAS scores at 0, 1, 3, 6, 12, 24 hours and 3th month after extubation. The VAS is an 11 point numeric scale which ranges from 0 to 10 at rest and during activity.
The number of patient requiring rescue analgesia | Postoperative day 1
  The number of patients who required rescue analgesics were recorded at 0, 1, 3, 6, 12 and 24. hours after extubation
Number of patients with postoperative nausea-vomiting and need of antiemetic usage | Postoperative day 1
  The severity of postoperative nausea and vomitting (PONV) was assessed using a descriptive verbal rating scale at 0, 1, 3, 6, 12 and 24 hours after extubation. If a score of 2 or more granisetron 1,5 mg iv will be administered. The PONV scale 0= no nausea, 1= slight nausea 2= moderate nausea, 3= vomiting once, 4= vomiting more than once
Remifentanil consumption during the surgery | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 160 min]
  The total amount of remifentanil consumed will be recorded.
Postoperative first oral intake time, first urination, first defecation time, first mobilization time, hospitalization time | Postoperative 7 days on an average
  Postoperative first oral intake time, first urination, first defecation time, first mobilization time, hospitalization time were recorded
Incidence of pruitus | Postoperative day 1
  Number of patient with pruitus were recorded at 0, 1, 3, 6, 12 and 24. hours

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Burcu Üstün, Prof, Study Director — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Özgenur Kekül, Samsun, Other, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, El-Boghdadly K. Mechanisms of action of the erector spinae plane (ESP) block: a narrative review. Can J Anaesth. 2021 Mar;68(3):387-408. doi: 10.1007/s12630-020-01875-2. Epub 2021 Jan 6. PMID 33403545
- [Background] Tulgar S, Selvi O, Senturk O, Serifsoy TE, Thomas DT. Ultrasound-guided Erector Spinae Plane Block: Indications, Complications, and Effects on Acute and Chronic Pain Based on a Single-center Experience. Cureus. 2019 Jan 2;11(1):e3815. doi: 10.7759/cureus.3815. PMID 30868029
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Kendall MC, Alves L, Traill LL, De Oliveira GS. The effect of ultrasound-guided erector spinae plane block on postsurgical pain: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 May 1;20(1):99. doi: 10.1186/s12871-020-01016-8. PMID 32357842